CLINICAL TRIAL: NCT00851604
Title: Evaluation of Serological Markers ProGRP, CgA, NSE and TUM2-PK in Patients With Malignant Neuroendocrine Tumors
Brief Title: ProGRP, CgA, NSE and TUM2-PK in in Patients With Neuroendocrine Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Asher Salmon, Hadassah Medical Organization
Other Study IDs: 052508-HMO-CTIL
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Neuroendocrine Tumors
Keywords: ProGRP; CgA; NSE; TUM2-PK; Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with malignant neuroendocrine tumors

SUMMARY:
The purpose of this study is to determine whether monitoring of levels of Serological Markers ProGRP, CgA, NSE and Pyruvate Kinase M2 are effective in the Evaluation of Diagnosis, Monitoring Therapeutic Effects and Predicting response to somatostatin analogues in Patients with Malignant Neuroendocrine Tumors.

DETAILED DESCRIPTION:
Assessment of the anatomical spread and disease progression in neuroendocrine tumor patients has become an essential part of disease management, but sometimes in many patients difficult to be measured. Therefore, the evaluation of serum markers could represent a useful tool for monitoring the course of the disease and the response of patients to therapy or palliative treatment.Clinical data considers CgA and NSE as available today blood biomarkers for neuroendocrine tumors.Until now the usefulness of serum ProGRP as a clinical tumor marker has been evaluated mainly in Small Cell Lung Carcinoma, while its role in the management of NE tumors has not been elucidated.Available in the literature limited data suggests that ProGRP may be a potential tumor marker in NE tumors.

Pyruvate kinase type M2 is the key glycolytic regulator in tumor cells.It catalyzes the dephosphorylation of phosphoenolpyruvate to pyruvate with ATP production.The dimeric form of this enzyme (TUM2-PK) has been detected in the blood of patients with different cancers.High TUM2-PK expression was suggested to be an important element of tumor cell metabolism adaptation to an inadequate oxygen and nutrient supply.Recently, it has been shown that somatostatin and its structural analogues pass through cell membrane and actively bind to cytosolic TUM2-PK. In response to this binding TUM2-PK translocates into the nucleus and induce programmed cell death. It is suggested that TUM2-PK enzyme may contribute significantly to response of neuroendocrine tumors to somatostatin analogues.

ELIGIBILITY:
Inclusion Criteria:

* The patients at diagnosis of neuroendocrine tumors before therapy will be approached to participate in the study.
* Older then 18 years old
* Patients who agree to participate will receive a detailed explanation and sign an informed consent form.

Exclusion Criteria:

* Pregnant women
* Coexistence of another primary malignant tumor other then neuroendocrine tumors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with neuroendocrine tumors
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Asher Salmon, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel